CLINICAL TRIAL: NCT00739869
Title: Effects of Hormone Therapy on Subclinical Neurological Pathology-The WHIMS-MRI Collaborative Study
Brief Title: Evaluating the Effects of Hormone Replacement Therapy on Brain Function (The WHIMS-MRI Study)
Acronym: WHIMS-MRI
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 571; N01-WH-4-4221
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: Silent Infarcts; Magnetic Resonance Imaging; MRI; Subclinical Cerebrovascular Disease; White Matter Grade Abnormalities; Total Brain Volume; Ventricular and Hippocampal Volume; Subclinical Vascular Abnormalities; Cerebrovascular Disease; CVD; Subclinical CVD
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Participants will include women who participated in the Women's Health Initiative Memory Study.

SUMMARY:
A silent stroke is a type of stroke that does not produce any severe symptoms, but may slightly affect memory or thinking abilities. Women who take hormone replacement therapy (HRT) may have a higher risk of experiencing a silent stroke than women who do not use HRT. This study will use magnetic resonance imaging (MRI) to determine the prevalence of silent strokes and other changes in brain tissue in women who participated in the Women's Health Initiative Memory Study (WHIMS), a study in which women received HRT, either as estrogen alone or as estrogen and progesterone combined, or placebo.

DETAILED DESCRIPTION:
A silent stroke is a type of stroke that occurs as a result of blockage in the small blood vessels in the brain. Older adults, in particular, are at risk for silent strokes. This type of stroke does not cause any of the typical stroke symptoms, such as vision problems, facial numbness, or walking difficulties; however, subtle changes in a person's cognitive ability or memory may occur following a silent stroke. It is important to diagnose this type of stroke because several occurrences of silent strokes can increase the risk of having a more serious, and possibly fatal, stroke. As women go through menopause, many choose to take HRT to relieve common menopausal symptoms, including hot flashes and mood swings. Unfortunately, the use of HRT may place women at higher risk of experiencing a silent stroke. This study will assess whether women who take HRT, either as estrogen alone or as estrogen and progesterone combined, have a greater risk of silent stroke than women who do not take HRT. Study researchers will also examine changes in brain tissue and changes in the areas of the brain associated with thinking and memory.

This study will enroll women who are participating in the WHIMS study. Participants will attend one study visit at which time a brain MRI scan will be completed. Study researchers will analyze participants' study data from the WHIMS study and the Women's Health Initiative Study of Cognitive Aging (WHISCA) study, an ancillary WHIMS study that examined the effects of HRT on memory and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the WHIMS study
* Receives medical care at 1 of the 13 WHIMS MRI clinics

Exclusion Criteria:

* Currently has a pacemaker (either working or non-functioning), intracranial aneurysm clip, neurostimulator, defibrillator, intra-ocular ferrous foreign body (e.g., metal in the eye), or Harrington rods
* Currently has a magnetically or electrically activated device, including any of the following items: cochlear implant, transcutaneous electrical nerve stimulation (TENS) unit, implanted pump (insulin or infusion), or a McGee Stapes implant
* Potential participants who have the following exclusion criteria may be eligible for participation, based on study staff approval:

  1. Metal fragments around critical soft tissue (i.e., shrapnel near spinal cord)
  2. Prosthetics
  3. Eyelid spring or wire
  4. Metallic stent, filter, or coil
  5. Breast tissue expander
  6. Tattoo or non-removable body piercing
  7. Difficulty lying flat
  8. Difficulty breathing
  9. Claustrophobia

Ages: 65 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Women who participated in the WHIMS study and receive medical care at clinics participating in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1426 (Actual)
Dates: Start 2004-05; Primary Completion 2006-04 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of silent infarcts in women assigned to HRT versus women assigned to placebo | Measured at a single study visit

CONTACTS AND LOCATIONS:
Overall Officials: Sally A. Shumaker, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Jaramillo SA, Felton D, Andrews L, Desiderio L, Hallarn RK, Jackson SD, Coker LH, Robinson JG, Ockene JK, Espeland MA; Women's Health Initiative Memory Study Research Group. Enrollment in a brain magnetic resonance study: results from the Women's Health Initiative Memory Study Magnetic Resonance Imaging Study (WHIMS-MRI). Acad Radiol. 2007 May;14(5):603-12. doi: 10.1016/j.acra.2007.02.001. PMID 17434074